CLINICAL TRIAL: NCT02302040
Title: mHealth Approach to Collaborative Asthma Management for Teens & Parents
Brief Title: Applying Interactive Mobile Health to Asthma Care in Teens (AIM2ACT)
Acronym: AIM2ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Miriam Hospital (Other); Rhode Island Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400921 - N; 1R21HD083830-01A1 (NIH)
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Asthma
Keywords: Adolescent
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIM2ACT (Experimental): AIM2ACT uses existing mHealth technology developed by the study team to elucidate tailored intervention targets for each family. AIM2ACT then facilitates collaborative caregiver/adolescent asthma management by automatically guiding dyads through a structured process that includes the supportive behavioral management strategies of goal setting, contingency management, and problem solving communication. Skills-training videos for adolescents and caregivers provide guidance on how to complete each collaborative asthma management component.
  Interventions: Behavioral: AIM2ACT
- Self-Guided (Active Comparator): Participants in the self-guided control condition will be given general information on supportive behavioral management techniques they can use to target improvement in asthma self-management behaviors. The control condition will serve as an attention control and is designed to optimize recruitment and sustain interest while concurrently having a minimal impact on asthma management.
  Interventions: Behavioral: Self-guided

INTERVENTIONS:
Behavioral: AIM2ACT — AIM2ACT is a mobile health tool that is designed to facilitate collaborative asthma management between early adolescents and their caregivers.
  Arms: AIM2ACT
Behavioral: Self-guided — Paper feedback and collaborative asthma management strategies are provided to early adolescents and caregivers.
  Arms: Self-Guided

SUMMARY:
The aims of this application are to develop and test AIM2ACT, a mobile health (mHealth) tool, delivered via smartphones, that fosters helpful caregiver support as early adolescents (ages 12-15) with persistent asthma develop and master asthma self-management behaviors. To facilitate helpful caregiver support, AIM2ACT uses mHealth technology to determine tailored intervention targets for each family. AIM2ACT then helps caregiver/adolescent dyads set asthma management goals by automatically guiding families through a structured process that includes the supportive behavioral management strategies of goal setting, contingency management, and problem solving communication. Skills-training videos for adolescents and caregivers provide guidance on how to complete each collaborative asthma management component.

AIM2ACT will be developed through feedback from an advisory board of adolescent-caregiver dyads from the target user population and a pediatric pulmonologist. Following advisory board feedback, the investigators will conduct a pilot randomized controlled trial of AIM2ACT with 50 early adolescents with poorly controlled asthma, ages 12-15 years, and a caregiver. Families will be randomly assigned to receive AIM2ACT or a self-guided condition for a 4 month intervention period. Participants in the self-guided condition will be given general information on supportive behavioral management techniques they can use to target improvement in asthma self-management behaviors. Outcomes include whether participants prefer AIM2ACT or the self-guided condition. Additionally, AIM2ACT and the self-guided condition will be compared to see if there are differences in changes in family asthma management (primary outcome), lung function, asthma control, asthma-related quality of life, and self-efficacy for asthma management. Data will be collected before participants are assigned to AIM2ACT or the self-guided control, post-treatment, and 4 month follow-up time points.

DETAILED DESCRIPTION:
As a participant in the study the following will take place:

Questionnaires will be filled out which will include medical history, including asthma symptoms and control, and questions related to quality of life. In addition, an interview will be completed which assesses the participants asthma management.

During this visit a brief training on how to complete lung function testing with a portable device will be demonstrated. The participant will breathe into twice per day for 14 days and then the device will be collected at the end of the 14 day period.

Randomization A computer will randomly chose one of the two programs; Program A or Program B. Random assignment is like rolling a dice to decide which group a person is assigned to. Both Program A and B are 4 months in length.

Program A the participant will answer questions about asthma management for a one-week period on a smartphone program. A smartphone can be provided for the duration of the study. After the one-week period, a report will be received on the smartphone about areas of asthma management that are going well and areas that may be in need of improvement. Next, brief meetings with study personnel to help determine things that will help improve asthma management. This information will be entered into a smartphone program. The participant will continue to use the smartphone program for a four month period.

Program B the participant answer questions about asthma for a one-week period on a paper and pencil diary. The participant will receive a paper copy of feedback from study personnel related to areas of asthma management that are going well and areas that may be in need of improvement. The participant will then be given information on techniques they can use to target identified areas for improvement. The participant will be encouraged to use these strategies to for a 4 month period.

ELIGIBILITY:
Inclusion Criteria:

* Lives in residence of caregiver,
* adolescent meets screening criteria for current persistent asthma,
* adolescent has uncontrolled asthma as indicated by a score of ≤ 19 on the Asthma Control Test,
* poorly controlled asthma according to National Heart, Lung, and Blood Institute (NHLBI) guidelines
* adolescent-caregiver dyad speak and read English

Exclusion Criteria:

* family is currently involved in an asthma management intervention, or
* adolescent has well controlled asthma as indicated by a score of ≥ 20 on the Asthma Control Test.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2015-12; Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Family asthma management system scale (FAMSS) will be measured for changes in baseline, 4 months, and 8 months. | Change in baseline, 4 months, and 8 months.
  Family Asthma Management System Scale (FAMSS) a validated family clinical interview that assesses core aspects of asthma management including medication adherence, symptom assessment and response, and integration of asthma into the family system.

SECONDARY OUTCOMES:
Spirometry will be used to measure a change in lung function at baseline, 4 months, and 8 months. | Change in baseline, 4 months, and 8 months.
  Lung function will be measured with spirometry at baseline, 4 months, and 8 months between the two groups to determine if the use of the AIM2ACT mHealth platform improved symptoms.
Asthma control test questionnaire will be used to measure a change in symptoms at baseline, 4 months, and 8 months. | Change in baseline, 4 months, and 8 months.
  Asthma control test questionnaire will be used to measure a change in symptoms at baseline, 4 months, and 8 months.
Asthma-related quality of life questionnaires will be given to measure the overall quality of life changes in baseline, 4 months, and 8 months.. | Change in baseline, 4 months, and 8 months.
  Asthma-related quality of life questionnaires will be given to measure the overall quality of life changes in baseline, 4 months, and 8 months.
Self-efficacy for asthma management questionnaire will be given to measure the overall improvement of the quality of life change in baseline, 4 months, and 8 months. | Change in baseline, 4 months, and 8 months.
  Asthma management efficacy questionnaire will be given to measure the overall improvement of the quality of life change in baseline, 4 months, and 8 months.
Family communication during asthma-management tasks will be assessed via the Decision Making Involvement Scale caregiver- and adolescent-reports at baseline and 4 months. | Change in baseline and 4 months
  Family communication during asthma-management tasks will be assessed via the Decision Making Involvement Scale caregiver- and adolescent-reports at baseline and 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: David A Fedele, Ph.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Benton Pediactrics, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fedele DA, Thomas JG, McConville A, McQuaid EL, Voorhees S, Janicke DM, Abu-Hasan M, Chi X, Gurka MJ. Using Mobile Health to Improve Asthma Self-Management in Early Adolescence: A Pilot Randomized Controlled Trial. J Adolesc Health. 2021 Dec;69(6):1032-1040. doi: 10.1016/j.jadohealth.2021.06.011. Epub 2021 Jul 15. PMID 34274211
- [Derived] Fedele DA, McConville A, Graham Thomas J, McQuaid EL, Janicke DM, Turner EM, Moon J, Abu-Hasan M. Applying Interactive Mobile health to Asthma Care in Teens (AIM2ACT): Development and design of a randomized controlled trial. Contemp Clin Trials. 2018 Jan;64:230-237. doi: 10.1016/j.cct.2017.09.007. Epub 2017 Oct 3. PMID 28986245